CLINICAL TRIAL: NCT05058664
Title: Developing Text-based Support for Parents of Suicidal Adolescents After Emergency Department Visits: A Multi-component Intervention Pilot
Brief Title: Developing Text-based Support for Parents of Adolescents After an Emergency Department Visit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ewa Czyz, Assistant Professor, Department of Psychiatry, University of Michigan, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HUM00184110; 1R34MH124767-01 (NIH)
Record Dates: First submitted 2021-09-16; First posted 2021-09-28 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Suicide
Keywords: Emergency Department
MeSH Terms: conditions — Suicide; Emergencies

STUDY DESIGN:
Intervention Model Description: There are 3 arms: control and 2 intervention arms. One of the intervention arms includes further twice daily (within-person) randomizations.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (standard care) (No Intervention)
- A-F texting component (Experimental): The A-F texting component will include content consistent with best-practice recommendations for parents to buffer youth against suicide risk.
  Interventions: Behavioral: A-F texting component
- A-F texting plus P-F texting component (Experimental): A-F texting plus P-F texting component arm includes the A-F component, as above, and P-F component. The P-F component includes an embedded micro-randomized trial (MRT) involving two daily randomizations to P-F message vs. no message conditions for the duration of the 6-week intervention. Participants who are randomized to this arm will be randomized twice each day (morning and evening) to either receive or not receive the P-F message at each randomization.
  Interventions: Behavioral: A-F texting component; Behavioral: P-F texting component

INTERVENTIONS:
Behavioral: A-F texting component — Over the course of the 6-week intervention parents in the A-F condition will receive 1 message each day.
  Arms: A-F texting component; A-F texting plus P-F texting component
Behavioral: P-F texting component — Over the course of the 6 week intervention, parents will receive between 1-2 messages, depending on randomization (in addition to A-F component messages)
  Arms: A-F texting plus P-F texting component

SUMMARY:
The researchers seek to develop a text message intervention for caregivers of adolescents at elevated suicide risk following discharge from emergency department (ED) care.

DETAILED DESCRIPTION:
Participants in the trial included 120 youth-parent dyads (120 youths and 120 parents). As the ultimate focus of the intervention is on improving youth outcomes, participant-related descriptives are provided for youth participants, except where noted specifically to be parent-related data.

ELIGIBILITY:
Parent eligibility:

Inclusion Criteria:

* Parent of eligible teen

Exclusion Criteria:

* Not owning a cell phone with text messaging capability.

Teen eligibility:

Inclusion Criteria:

* Recent suicidal ideation (within last 2 weeks) and/or suicide attempt within the last month.

Exclusion Criteria:

* Youth with severe cognitive impairment or altered mental status (e.g., psychosis, manic state)
* Youth with severe aggression/agitation
* No availability of a legal guardian

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Czyz, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Czyz E, Nahum-Shani I, Ewell Foster C, Micol V, Jiang A, Al-Dajani N, Arango A, Walton M, Hong V, Ahamed SI, King C. Building toward a text-based intervention for parents of suicidal adolescents seeking emergency department care: A pilot randomized controlled trial. J Consult Clin Psychol. 2025 May;93(5):382-389. doi: 10.1037/ccp0000950. PMID 40354273

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Unless indicated otherwise, the data shown below represent youth participants, as they were the object of the study.
  Of 125 youth participants consented, 5 were removed due to administrative issues. 4 participants were not randomized due to a platform glitch, and 1 consented participant turned out to be ineligible. These 5 were not included in the analysis, so 120 dyads are included in the trial.
Groups:
- Control (Standard Care): Standard Emergency Department services (usual care)
Period: Overall Study
Arm/Group | Control (Standard Care) | A-F Texting Component | A-F Texting Plus P-F Texting Component
Started (Participant numbers shown represent dyads of one adolescent and one caregiver.) | 37 | 42 | 41
Completed | 33 | 42 | 38
Not Completed | 4 | 0 | 3
Not completed — No follow-up data provided | 4 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Standard Care) | A-F Texting Component | A-F Texting Plus P-F Texting Component | Total
Number analyzed (Participants) | 37 | 42 | 41 | 120
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age of adolescent members of dyads | 15.03 (1.42) | 14.55 (1.43) | 14.98 (1.19) | 14.84 (1.36)
  Age of caregiver members of dyads | 45.03 (8.15) | 43.74 (5.89) | 45.20 (6.15) | 44.63 (6.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex of adolescent members of dyads: Female | 23 | 29 | 27 | 79
  Sex of adolescent members of dyads: Male | 14 | 13 | 14 | 41
  Sex of caregiver members of dyads: Female | 31 | 38 | 37 | 106
  Sex of caregiver members of dyads: Male | 6 | 4 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity of adolescent members of dyads: Hispanic or Latino | 4 | 2 | 3 | 9
  Ethnicity of adolescent members of dyads: Not Hispanic or Latino | 28 | 36 | 32 | 96
  Ethnicity of adolescent members of dyads: Unknown or Not Reported | 5 | 4 | 6 | 15
  Ethnicity of caregiver members of dyads (not collected): Hispanic or Latino | 0 | 0 | 0 | 0
  Ethnicity of caregiver members of dyads (not collected): Not Hispanic or Latino | 0 | 0 | 0 | 0
  Ethnicity of caregiver members of dyads (not collected): Unknown or Not Reported | 37 | 42 | 41 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race of adolescent members of dyads: American Indian or Alaska Native | 1 | 0 | 1 | 2
  Race of adolescent members of dyads: Asian | 1 | 0 | 1 | 2
  Race of adolescent members of dyads: Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  Race of adolescent members of dyads: Black or African American | 2 | 4 | 3 | 9
  Race of adolescent members of dyads: White | 25 | 34 | 31 | 90
  Race of adolescent members of dyads: More than one race | 4 | 4 | 1 | 9
  Race of adolescent members of dyads: Unknown or Not Reported | 2 | 0 | 4 | 6
  Race of caregiver members of dyads: American Indian or Alaska Native | 0 | 1 | 0 | 1
  Race of caregiver members of dyads: Asian | 2 | 0 | 1 | 3
  Race of caregiver members of dyads: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race of caregiver members of dyads: Black or African American | 2 | 2 | 2 | 6
  Race of caregiver members of dyads: White | 32 | 38 | 37 | 107
  Race of caregiver members of dyads: More than one race | 1 | 0 | 1 | 2
  Race of caregiver members of dyads: Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: dyads]
  United States | 37 | 42 | 41 | 120

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eligible Youth-Parent Dyads Who Agree to Participate in the Study,
Description: Data represent participant dyads who were eligible and approached about study participation, and who agreed to take part in the study.
Time Frame: At the time of youth Emergency Department visit
Population: The data shown here represent potential youth participants who were eligible, as indicators of the dyad because they were the focus of the study.
Measure: Count of Units; unit: Parent-youth dyads
Units Other Than Participants: Parent-youth dyads
Groups:
- Participants Consented: Eligible individuals who were approached about study participation and who agreed to take part in the study
Arm/Group | Participants Consented
Number analyzed (Participants) | 207
Number analyzed (Parent-youth dyads) | 207
Parent-youth dyads | 125

2. Primary Outcome: Participant Dyads Who Completed Follow-up Assessments
Description: Data was used to determine retention rate among the participant dyads. We report on follow up completion for both adolescent and caregiver members of the dyad.
Time Frame: Up to 12 weeks
Measure: Count of Units; unit: Responses from dyad members
Units Other Than Participants: Responses from dyad members
Groups:
- Control: Standard care
Arm/Group | Control | A-F Texting Component | A-F Texting Plus P-F Texting Component
Number analyzed (Participants) | 37 | 42 | 41
Number analyzed (Responses from dyad members) | 37 | 42 | 41
Responses from dyad members
  Count of Parent responses | 33 | 42 | 38
  Count of Adolescent Responses | 29 | 35 | 27

3. Primary Outcome: Percentage of Participants Randomized to the Intervention Who Remained Active (Texting Arms Only)
Description: Results represent parent participants who did not request stopping the intervention (i.e., did not request to stop receiving messages).
Time Frame: Up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | A-F Texting Component | A-F Texting Plus P-F Texting Component
Number analyzed (Participants) | 42 | 41
Participants | 42 | 39

4. Primary Outcome: Participating Parents' Satisfaction With the Intervention (Texting Arms Only)
Description: Measured using the Modified Client Satisfaction Questionnaire (CSQ), which was a 2-question survey. Each question had a range of 1-4. Adult participants were asked to rate both their overall satisfaction (1 meaning not satisfied to 4 meaning highly satisfied), and the likelihood that they would recommend their particular assigned intervention to a friend (1 meaning highly unlikely to 4 meaning highly likely).
Time Frame: Up to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-F Texting Component | A-F Texting Plus P-F Texting Component
Number analyzed (Participants) | 39 | 35
score on a scale
  Overall satisfaction | 3.51 (0.56) | 3.37 (0.60)
  Recommend to a friend | 3.56 (0.55) | 3.43 (0.66)

5. Primary Outcome: Number of and Reasons for Active Withdrawals
Description: Parent participant request to withdraw from the study. Study intention was to collect the number of and reasons for withdrawals, but the sole withdrawal did not provide a reason.
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | A-F Texting Component | A-F Texting Plus P-F Texting Component
Number analyzed (Participants) | 37 | 39 | 35
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Description: Since all youth participants were enrolled because of emergency dept. visit for suicide risk (ideation or attempts), those who were unreachable at follow-up were not included in denominators of suicide attempts, as they could not be presumed to have or not to have attempted suicide. Thus it is most accurate to report only known data that is based on collected AEs. Non-serious Adverse Events were not collected.
  Deaths and Adverse Events were not assessed/monitored in Parents.
Arm/Group | Control | A-F Texting Component | A-F Texting Plus P-F Texting Component
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 5/21 | 2/26 | 1/23
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=21) | A-F Texting Component (N=26) | A-F Texting Plus P-F Texting Component (N=23)
Suicide attempt (Psychiatric disorders) | 5 | 2 | 1 — As noted above, those who were unreachable at follow-up were not included in denominators of suicide attempts, as they could not be presumed to have or not to have attempted suicide.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT05058664/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/64/NCT05058664/ICF_000.pdf